CLINICAL TRIAL: NCT05039437
Title: Development of Green Mei Products for the Prevention of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS2-19033
Record Dates: First submitted 2021-08-12; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MGF-4 (Experimental): Take two MGF-4 capsules twice a day for 8 weeks. A 250 mg capsule contents 243 mg MGF-4 and other excipients.
  Interventions: Dietary Supplement: MGF-4
- MGF-7 (Experimental): Take two MGF-7 capsules twice a day for 8 weeks. A 250 mg capsule contents 243 mg MGF-7 and other excipients.
  Interventions: Dietary Supplement: MGF-7

INTERVENTIONS:
Dietary Supplement: MGF-4 — Participants were instructed to take 2 capsules of MGF-4 twice a day, and measure own blood pressure at morning everyday throughout the duration of the study.
  Arms: MGF-4
Dietary Supplement: MGF-7 — Participants were instructed to take 2 capsules of MGF-7 twice a day, and measure own blood pressure at morning everyday throughout the duration of the study.
  Arms: MGF-7

SUMMARY:
The aim of this study is to investigate the antihypertensive effects of Mei-Gin formula-4 (MGF-4) and Mei-Gin formula-7.

DETAILED DESCRIPTION:
It's a randomized, and single-blind trial and was designed to evaluate the effects of MGFs (MGF-4 and MGF-4) on blood pressure. 50 participants with hypertension (systolic blood pressure between 130-179 mmHg or diastolic blood pressure between 85-109 mmHg) who did not accept any hypertension medication were randomized allocated to either MGF-4 or MGF-7 group. Participants were instructed to take 4 capsules of MGF-4 or MGF-7 daily throughout the duration of the 8 weeks intervention study. After treatment, the change of the blood pressure and relative mechanism were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The age of the subject is 20 to 70 years old.
* The subject is a patient with hypertension (SBP is between 130-179 mmHg, DBP is between 85-109mmHg, one of the two can be diagnosed), and there are no serious illnesses requiring hospitalization during the study period treatment.
* No hypertension medication.
* The subject can understand the test process described in the consent form and the possible potential risks and benefits, and able to sign the consent form.
* The subjects shall observe diet control during the trial period.

Exclusion Criteria:

* Subjects diagnosed with cancer and still under active treatment.
* Subjects diagnosed with heart disease and still under active treatment.
* Other drugs are used, whose pharmacological effects may affect blood pressure or may aggravate the effects of drugs.
* Subjects who have systemic infection and need systemic antibiotics.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change the blood pressure after intervention | Week 0, 4 and 8
  Compare the difference of own SBP and DBP between the week 0, 4 and 8 in each groups

SECONDARY OUTCOMES:
Change from baseline serum MDA and TEAC at Week 8 | Week 0 and 8
  Compare the difference of serum MDA and TEAC between week 0 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Han-Hui Chang, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan